CLINICAL TRIAL: NCT04472611
Title: Colchicine/Statins for the Prevention of COVID-19 Complications (COLSTAT) Trial
Acronym: COLSTAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000027950
Record Dates: First submitted 2020-07-14; First posted 2020-07-15 (Actual); Results first posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: SARS-CoV-2
Keywords: Rosuvastatin; Colchicine
MeSH Terms: interventions — Standard of Care; Colchicine; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care (SOC) and Colchicine+Rosuvastatin (Experimental): Patients will take Rosuvastatin 40mg daily and Colchicine 0.6mg twice for 3 days and then 0.6mg daily during hospitalization
  Interventions: Drug: Standard of Care (SOC) and Colchicine+Rosuvastatin
- Standard of care (SOC) (No Intervention): Patients will undergo standard of care treatment during hospitalization determined by the primary care team during hospitalization

INTERVENTIONS:
Drug: Standard of Care (SOC) and Colchicine+Rosuvastatin — Patients will take Rosuvastatin 40mg daily and Colchicine 0.6mg twice for 3 days and then 0.6mg daily during hospitalization
  Other Names: SOC & Colchicine and Rosuvastatin
  Arms: Standard of Care (SOC) and Colchicine+Rosuvastatin

SUMMARY:
This is a pragmatic randomized open-label study of the safety and efficacy of the combination of colchicine and Rosuvastatin in addition to standard of care (SOC) compared to SOC alone in hospitalized patients with SARS-CoV-2

DETAILED DESCRIPTION:
This is a prospective 1:1 randomized open-label clinical trial to investigate the safety and efficacy of the combination of Colchicine + Rosuvastatin added to standard of care (SOC) compared to SOC alone in hospitalized subjects with moderate COVID-19.

Subjects will be screened during admission to hospital. Patients with confirmed SARS-CoV-2 infection, and meeting all other inclusion and exclusion criteria, will be randomized to either Colchicine+Rosuvastatin treatment or SOC for the duration of hospitalization. SOC will be guided by the YNHH SARS-CoV-2 Therapeutics Group. In cases where patients require randomization in another trial evaluating an experimental drug, they will continue on study drug. Patients will be assessed daily while hospitalized for clinical, biomarker, safety, and laboratory parameters based on SOC.

Colchicine is an extensively studied oral anti-inflammatory agent with a well-defined safety profile. Colchicine, by inhibiting tubulin polymerization and clathrin-mediated endocytosis has the potential to inhibit SARS-CoV-2 cell entry. In addition, colchicine has a direct anti-inflammatory effect by inhibiting the NLRP3 inflammasome activation which in turn has the potential to reduce the SARS-CoV-2-induced cytokine storm. Statins also have direct anti-inflammatory effects by reducing chemokine release, adhesion molecules, and modulating T cell activity and have the potential to prevent SARS-CoV-2 related endothelial dysfunction and may reduce the morbidity and mortality associated with COVID-19. Rosuvastatin, in particular, appears to have direct antiviral properties by binding and inhibiting the active site of the main protease enzyme (Mpro) of SARS-CoV-2.1

The combination Colchicine + Rosuvastatin may have a synergetic effect to antagonize SARS-CoV-2 infection, modulate the inflammatory response and to reduce morbidity and mortality associated with acute respiratory distress syndrome (ARDS) and myocardial injury in COVID-19 patients.

Both drugs have been in use for decades for gout and pericarditis (colchicine) and hyperlipidemia, coronary disease (CAD) and diabetes (rosuvastatin/Crestor), and have been tested in thousands of patients used individually and in combination with a low and well characterized risk profile. Colchicine and rosuvastatin are currently used as standard of care in COVID-19 patients whether due to pre-existing CAD, gout or pericarditis or acute presentations with acute coronary syndromes or acute gout with no expected added risk in the population being studied.

This study is not intended to support a labeling change or advertising claim for either drug, and the study will be conducted in compliance with the requirements of Yale University's IRB review and a research IND.

Subjects will be screened within 48 hours of hospital admission. Patients with real-time reverse transcription polymerase chain reaction (RT-PCR) confirmed SARS-CoV-2 infection and meeting all inclusion and exclusion criteria, will be randomized to either Colchicine + Rosuvastatin treatment in addition to SOC or SOC alone for the duration of hospitalization.

Subjects will be randomized in a 1:1 manner to one of two arms:

Active treatment:

In addition to SOC* subjects randomized to active treatment will receive:

* Rosuvastatin: 40mg daily AND
* Colchicine: 0.6mg twice daily for 3 days then 0.6mg daily Note: Dose adjustment based on medical conditions and drug interactions (see section §7.4.1). Subjects previously on chronic statin therapy will be eligible for enrollment in the trial, and if randomized to active treatment, chronic statin therapy will be discontinued and replaced by rosuvastatin 40 mg for 30 days or hospital discharge and resumed thereafter.

Standard of Care Controls:

Subjects will undergo SOC treatment determined by the primary care team and the YNHH treatment algorithm for hospitalized patients with COVID-19.

*All standard of care treatments for hospitalized subjects with SARS-CoV-2 are permitted concurrently with the study intervention. This only includes treatments approved by the Yale SOC treatment Committee. Concomitant therapy will be performed according to standard practice, local standards of care and published guidelines. Subjects will not be permitted to participate in other investigational studies. Methods for identifying drug interactions and dose adjustment are listed in section §7.4.1 of the protocol. Drug discontinuation is only permitted with documented adverse reactions (section §7.4.3).

Treatment will continue for a total of 30 days. If the subject is discharged the treatment will stop at that time.

ELIGIBILITY:
Inclusion Criteria 1.18 years or older and confirmed SARS-CoV-2 infection by RT-PCR 2. Patient is admitted to the floor (non-ICU) within 48 hours of hospital admission 3. The patient, or legally authorized representative, has been informed of the nature of the study, agrees to its provisions and has provided witnessed (by 2 independent members of the health care team) oral informed consent, or a photograph of the signed informed consent approved by the Institutional Review Board (IRB)

Exclusion Criteria:

1. Known pregnancy or nursing mothers
2. Known allergy to statins or colchicine
3. Patient is on chronic colchicine or oral corticosteroid treatment
4. Acute liver disease defined by elevated transaminases (AST/ALT > 3x ULN)
5. Severe chronic kidney disease defined as glomerular filtration rate (GFR) < 30mL/min1.73 m2
6. Severe QTc prolongation (>500ms narrow QRS<120ms and >550ms for wide QRS>120)
7. Presents with severe disease on admission (WHO ordinal scale of clinical improvement scores 5-8)
8. Rhabdomyolysis or CPK > 5x ULN
9. Thrombocytopenia defined as platelet count < 50,000 / mm3
10. Leukopenia defined as white blood cell count < 3000 ml
11. Severe anemia defined as Hemoglobin value <8 g/100ml
12. Participation in any other clinical trial of an experimental treatment for COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Lansky, MD, Principal Investigator — Yale University
Locations (4):
- United States (4):
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Greenwich Hospital, Greenwich, Connecticut
  - Yale New Haven Hosptial System, New Haven, Connecticut
  - Lawrence & Memorial Hospital, New London, Connecticut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shah T, McCarthy M, Nasir I, Archer H, Ragheb E, Kluger J, Kashyap N, Paredes C, Patel P, Lu J, Kandel P, Song C, Khan M, Huang H, Ul Haq F, Ahmad R, Howes C, Cambi B, Lancaster G, Cleman M, Dela Cruz C, Parise H, Lansky A. Colchicine and high-intensity rosuvastatin in the treatment of non-critically ill patients hospitalised with COVID-19: a randomised clinical trial. BMJ Open. 2023 Feb 24;13(2):e067910. doi: 10.1136/bmjopen-2022-067910. PMID 36828654
- [Derived] Shah T, McCarthy M, Nasir I, Archer H, Ragheb E, Kluger J, Kashyap N, Paredes C, Patel P, Lu J, Kandel P, Song C, Khan M, Ul Haq F, Ahmad R, Howes C, Cambi B, Lancaster G, Cleman M, Dela Cruz CS, Parise H, Lansky A. Design and rationale of the colchicine/statin for the prevention of COVID-19 complications (COLSTAT) trial. Contemp Clin Trials. 2021 Nov;110:106547. doi: 10.1016/j.cct.2021.106547. Epub 2021 Aug 28. PMID 34461322

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care (SOC) and Colchicine+Rosuvastatin | Standard of Care (SOC)
Started | 125 | 125
Completed | 122 | 125
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Population: Patients hospitalized with moderate to severe symptoms of COVID being treated with standard protocol medications as set by hospital
Groups:
- SOC and Colchicine and Rosuvastatin: Patients will take Rosuvastatin 40mg daily and Colchicine 0.6mg twice for 3 days and then 0.6mg daily during hospitalization
- Total: Total of all reporting groups
Arm/Group | SOC and Colchicine and Rosuvastatin | Standard of Care (SOC) | Total
Number analyzed (Participants) | 125 | 125 | 250
Age, Categorical [Count of Participants; unit: Participants] — Age 18+ hospitalized with COVID No liver, kidney issues
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 74 | 77 | 151
    >=65 years | 51 | 48 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (14.6) | 62.4 (16.1) | 61.4 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 55 | 124
  Male | 56 | 70 | 126
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 24 | 13 | 37
  White | 76 | 81 | 157
  More than one race | 24 | 27 | 51
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 125 | 125 | 250

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With COVID 19 Severity
Description: As defined by World Health Organization Ordinal Scale, which ranges from 1 to 8. Severity of COVID measured by WHO Scores 5-8: Defined as 5= Hospitalized requiring including CPAP, face mask, high flow nasal cannula (Excludes regular nasal cannula), 6= Hospitalized requiring intubation and mechanical ventilation, 7= Hospitalized requiring mechanical ventilation and additional organ support (vasopressors, renal replacement therapy, ECMO), 8= Death. Data presented is for Max WHO scores 5-8, indicating moderately to severely infected participants.
Time Frame: 30 Days
Population: Moderately infected COVID patients requiring hospitalization.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SOC) and Colchicine+Rosuvastatin | Standard of Care (SOC)
Number analyzed (Participants) | 17 | 8
Participants
  Max WHO score 5 | 5 | 4
  Max WHO score 6 | 2 | 0
  Max WHO score 7 | 4 | 1
  Max WHO score 8 | 6 | 3

ADVERSE EVENTS:
Time Frame: Adverse events were recorded for patients starting at date/time of enrollment through study exit at 60 day post-discharge timepoint.
Description: Adverse events were recorded for patients starting at date/time of enrollment through study exit at 60 day post-discharge timepoint, up to a maximum of 90 days.
Arm/Group | Standard of Care (SOC) and Colchicine+Rosuvastatin | Standard of Care (SOC)
All-Cause Mortality (participants affected / at risk) | 7/125 | 4/125
Serious Adverse Events (participants affected / at risk) | 4/125 | 4/125
Other Adverse Events (participants affected / at risk) | 9/125 | 2/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (SOC) and Colchicine+Rosuvastatin (N=125) | Standard of Care (SOC) (N=125)
Death (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4) — Respiratory failure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (SOC) and Colchicine+Rosuvastatin (N=125) | Standard of Care (SOC) (N=125)
Gastrointestinal Distress (Gastrointestinal disorders) | 5 (5) | 0 (0) — Diarrhea
Increased Liver Function Tests (Immune system disorders) | 4 (4) | 2 (2) — Increased amount of liver function test values

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-08): https://cdn.clinicaltrials.gov/large-docs/11/NCT04472611/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-06): https://cdn.clinicaltrials.gov/large-docs/11/NCT04472611/ICF_001.pdf